CLINICAL TRIAL: NCT03133455
Title: Repetitive Thoughts in Fibromyalgia: Impact of Rumination on the Emotional and Cognitive Dimensions of Fibromyalgia
Acronym: PRFM-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2015_843_0024
Record Dates: First submitted 2017-04-04; First posted 2017-04-28 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Fibromyalgia
Keywords: Rumination
MeSH Terms: conditions — Fibromyalgia; Rumination Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with Fibromyalgia (Other)
  Interventions: Other: Evaluate the link between an abstract / analytical thinking style and depressive manifestations in FM.

INTERVENTIONS:
Other: Evaluate the link between an abstract / analytical thinking style and depressive manifestations in FM. — Evaluate the link between an abstract / analytical thinking style and depressive manifestations in FM.

SUMMARY:
Dysfunctional chronic diffuse pain syndrome, concerning 2% of the French population, Fibromyalgia (FM) is classified either as a psychological disease or as a somatic disease. This dichotomous reasoning does not lead to a better understanding and does not allow the use or development of new psychological tools of care.

The issue of the proximity between FM and depression highlighted by some authors and the presence of anxious comorbidities may arise at a different level, that of the transdiagnostic approach. Rumination is one of these transdiagnostic processes that are the subject of recent studies and one of the dimensions of which (abstract analytical rumination) is at work in depression and a number of psychopathologies. The investigator therefore wishes to explore the process of rumination and its abstract analytical dimension in FM and to explore its link with the depressive and anxious manifestations frequently associated with this disorder.

ELIGIBILITY:
Inclusion Criteria:

* FM Criteria of the American College of Rheumatology ACR 1990.
* Major Patients
* free and informed consent signed
* stable treatment for at least one month
* Native French speaker
* Patient covered by health insurance.

Exclusion Criteria:

* Patient deprived of liberty or protected major (under guardianship or curatorship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2015-09-16 (Actual); Primary Completion 2017-11-26 (Actual); Study Completion 2017-11-26 (Actual)

PRIMARY OUTCOMES:
Analyze the rate of rumination and depression of a fibromyalgia patient using a questionnaire | 1 hour
  Analyze the rate of rumination and depression of a fibromyalgia patient using a questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France

REFERENCES:
- [Result] Fonseca Das Neves J, Serra E, Kosinski T, Marechal V, Rollin N, Richard O, Jehel L, Rusinek S. Catastrophizing and rumination mediate the link between functional disabilities and anxiety/depression in fibromyalgia. A double-mediation model. Encephale. 2024 Apr;50(2):162-169. doi: 10.1016/j.encep.2023.04.004. Epub 2023 May 1. PMID 37137739